CLINICAL TRIAL: NCT04075396
Title: A Phase I/II, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-Tumor Activity of YH25448 in Patients With EGFR Mutation Positive Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Lazertinib in Participants With Epidermal Growth Factor Receptor (EGFR) Mutation Positive Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108680; 73841937NSC2001 (Other: Janssen Research & Development, LLC); YH25448-201 (Other: Yuhan Corporation); 2019-003106-28 (EudraCT Number)
Record Dates: First submitted 2019-08-21; First posted 2019-08-30 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part D: Outside of Korea (Experimental): Participants from outside of Korea with progressive disease and on prior epidermal growth factor receptor (EGFR) Tyrosine kinase inhibitor (TKI) therapy will receive recommended phase 2 doses based on safety, tolerability, efficacy and pharmacokinetics (PK) of Lazertinib.
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib — Participants will receive Lazertinib tablets once daily.
  Other Names: YH25448; JNJ-73841937

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of Lazertinib when given orally to participants with epidermal growth factor receptor single activating mutation positive (EGFRm+) locally advanced or metastatic Non Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
One-third of all cancer deaths worldwide are still caused by lung cancer and non-small-cell lung cancer (NSCLC). Lazertinib is an oral, highly potent, mutant-selective and irreversible epidermal growth factor receptor (EGFR) Tyrosine kinase inhibitor (TKIs) targets both the T790M mutation and activating EGFR mutations while sparing wild type-EGFR. The study will be conducted in participants with EGFR mutation positive advanced non-small cell lung cancer (NSCLC). Study Parts A, B, and C are sponsored by Yuhan Corporation under protocol identifier YH25448-201 (ClinicalTrials.gov Identifier: NCT03046992), and Study Part D is sponsored by Janssen Research and Development, LLC under protocol identifier 73841937NSC2001. In Part D, Lazertinib will be given to participants outside Korea, including Caucasians, in order to evaluate safety, tolerability, efficacy (including tumor response) and Pharmacokinetics (PK) in participants outside of Korea. The duration of this study will be up to 2 years. Study treatment should be held in all participants with suspected (symptomatic) or documented severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) positive disease, until recovery from all infection related symptoms, and documented to be negative for SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Females should agree to use adequate contraceptive measure, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of following criteria at screening; Post-menopausal defined as aged more than 50 years and ameorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments; Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation; Women under 50 years old would be considered postmenopausal if they have been ameorrhoeic for at least 12 months following cessation of exogenous hormonal treatment, and have serum follicle-stimulating hormone (FSH) and luteinizing hormone (LH) levels in postmenopausal range for the institution
* Male participants who have not undergone a vasectomy must agree to use barrier contraception that is, condoms, and refrain from donating sperm until 3 months after last drug is taken
* During the study, and for 3 months after receiving the last dose of study drug, female participants must agree not to donate eggs (ova, oocytes) and male participants must agree not to donate sperm for the purposes of assisted reproduction
* In Part D: Participants outside Korea with histologically or cytologically (that is, using pleural effusion, ascites) confirmed Non-Small Cell Lung Cancer (NSCLC) with previously diagnosed epidermal growth factor receptor single activating mutation positive (EGFRm+), and who have had progressive disease on prior epidermal growth factor receptor- Tyrosine kinase inhibitor (EGFR-TKI) therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 3 months

Exclusion Criteria:

* An unapproved investigational product from another clinical study within 30 days of the first dose of study treatment
* Treatment with an EGFR TKIs (example: erlotinib or gefitinib) within 8 days or approximately 5x half-life, whichever is the longer, of the first dose of study treatment or other investigational products within approved indication of marketed product (if sufficient wash-out time has not occurred due to schedule or PK properties, an alternative appropriate wash-out time based on known duration of time to reversibility of drug related adverse events could be agreed upon by sponsor and the Investigator)
* Any cytotoxic chemotherapy or other anticancer drugs for the treatment of advanced NSCLC from a previous treatment regimen within 14 days of the first dose of study treatment
* Symptomatic spinal cord compression (if steroid treatment is not required within at least 2 weeks prior to the start of the study treatment then the participant may be enrolled)
* Brain metastases with symptomatic and/or requiring emergency treatment (example; Steroid for at least 2 weeks prior to start of study treatment)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (9):
- United States (5):
  - City of Hope, Duarte, California
  - Advent Health Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Montefiore Medical Center, The Bronx, New York
  - Tennessee Oncology, Nashville, Tennessee
- Spain (3):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp Virgen de La Victoria, Málaga
- The Christie Nhs Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Kim B, Lee J, Jang H, Lee N, Mehta J, Jang SB. Effects of Acid-Reducing Agents on the Pharmacokinetics of Lazertinib in Patients with EGFR Mutation-Positive Advanced Non-Small-Cell Lung Cancer. Adv Ther. 2022 Oct;39(10):4757-4771. doi: 10.1007/s12325-022-02286-z. Epub 2022 Aug 13. PMID 35962934

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Parts A, B, and C were sponsored by Yuhan Corporation under protocol identifier (ID) YH25448-201 and Part D was sponsored by Janssen Research and Development, LLC under protocol ID 73841937NSC2001. Therefore, only Part D results are reported.
Groups:
- Lazertinib (YH25448-201/JNJ-73841937) 240 mg: Participants with epidermal growth factor receptor single activating mutation positive (EGFRm+) advanced non-small cell lung cancer (NSCLC) with or without asymptomatic brain metastasis received lazertinib tablet at a dose of 240 milligrams (mg) orally on Day 1 of Cycle 0, which spans 7 days, followed by a once daily dose in each subsequent 21-day treatment cycle, for a maximum duration of up to 32.7 months. Participants were then followed up for safety for 28 days after the last dose of study treatment.
- Lazertinib 320 mg: Participants with EGFRm+ advanced NSCLC with or without asymptomatic brain metastasis received lazertinib tablet at a dose of 320 mg orally on Day 1 of Cycle 0, which spans 7 days, followed by a once daily dose in each subsequent 21-day treatment cycle, for a maximum duration of up to 8.3 months. Participants were then followed up for safety for 28 days after the last dose of study treatment.
Period: Overall Study
Arm/Group | Lazertinib (YH25448-201/JNJ-73841937) 240 mg | Lazertinib 320 mg
Started | 15 | 14
Treated (Safety Analysis Population) | 15 | 13
Completed | 0 | 0
Not Completed | 15 | 14
Not completed — Death | 11 | 9
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Participants did not complete the 28 days follow-up after implementation of protocol amendment 11 | 3 | 2
Not completed — Enrolled but not-treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis population included all participants who received at least 1 dose of investigational product (IP).
Groups:
- Lazertinib 240 mg: Participants with EGFRm+ advanced NSCLC with or without asymptomatic brain metastasis received lazertinib tablet at a dose of 240 mg orally on Day 1 of Cycle 0, which spans 7 days, followed by a once daily dose in each subsequent 21-day treatment cycle, for a maximum duration of up to 32.7 months. Participants were then followed up for safety for 28 days after the last dose of study treatment.
- Total: Total of all reporting groups
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (11.35) | 63 (12.48) | 61.7 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  SPAIN | 10 | 8 | 18
  UNITED KINGDOM | 0 | 1 | 1
  UNITED STATES | 5 | 4 | 9
Number of prior lines of therapy [Count of Participants; unit: Participants]
  <= 4 Lines | 8 | 4 | 12
  > 4 Lines | 7 | 9 | 16
Weight group [Count of Participants; unit: Participants]
  < 80 kilograms (kg) | 13 | 10 | 23
  >= 80 kg | 2 | 2 | 4
  Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part D: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs were defined as AEs that started on or after the first dose of study medication and prior to 28-day follow-up period. All TEAEs including serious and non-serious events are reported in this outcome measure.
Time Frame: From Day 1 up to 14 months
Population: The safety analysis population included all participants who received at least 1 dose of investigational product (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 15 | 13
Participants | 15 | 13

2. Primary Outcome: Part D: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Number of participants with clinically significant abnormalities in vital signs were reported. Vital signs included pulse rate, systolic blood pressure, diastolic blood pressure, body temperature, height, weight, and body mass index (BMI). Baseline was defined as last non-missing measurement taken prior to reference start date.
Time Frame: From Day 1 up to 14 months
Population: The safety analysis population included all participants who received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 15 | 13
Participants | 0 | 0

3. Primary Outcome: Part D: Number of Participants With Clinically Significant Abnormalities in Physical Examination
Description: Number of participants with clinically significant abnormalities in physical examination were reported. Physical examination included general appearance, skin, head and neck (including ears, eyes, nose and throat), respiratory, cardiovascular, abdomen, lymph nodes, thyroid, muscular-skeletal (including spine and extremities) and neurological systems. Baseline was defined as last non-missing measurement taken prior to reference start date.
Time Frame: From Day 1 up to 14 months
Population: The safety analysis population included all participants who received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 15 | 13
Participants | 8 | 2

4. Primary Outcome: Part D: Number of Participants With Greater Than or Equal to (>=) Grade 4 Toxicity in Laboratory Tests Based on National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version (v) 4.03
Description: Safety laboratory assessments included clinical chemistry, hematology and urinalysis. Grading was done as per NCI CTCAE version 4.03: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death. Baseline was defined as last non-missing measurement taken prior to reference start date.
Time Frame: From Day 1 up to 14 months
Population: The safety analysis population included all participants who received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 15 | 13
Participants | 2 | 0

5. Primary Outcome: Part D: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Tests
Description: Number of participants with clinically significant abnormalities in electrocardiogram (ECG) tests were reported. ECG variables included heart rate, PR interval, RR interval, QRS interval, QT interval and Fridericia-corrected QT interval (QTcF). Baseline was defined as last non-missing measurement taken prior to reference start date.
Time Frame: From Day 1 up to 14 months
Population: The safety analysis population included all participants who received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 15 | 13
Participants | 1 | 1

6. Primary Outcome: Part D: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-last]) for Single Dose of Lazertinib
Description: AUC(0-last) was defined as area under the plasma concentration-time curve from time zero to time of last quantifiable concentration. AUC(0-last) for single dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive liquid chromatography-mass spectrometry/mass spectrometry (LC-MS/MS) method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: Pharmacokinetic (PK) analysis population included all participants who had at least 1 measurable concentration collected post dose. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Hour*nanograms per milliliter (h*ng/mL)
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
Hour*nanograms per milliliter (h*ng/mL) | 5907.56 (2218.84) [lower limit 2218.84] | 7664.99 (2057.13) [lower limit 2057.13]

7. Primary Outcome: Part D: Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC[0-Infinity]) for Single Dose of Lazertinib
Description: AUC(0-infinity) was defined as area under the plasma concentration time curve from time zero to infinite time. AUC(0-infinity) for single dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: PK analysis population included all participants who had at least 1 measurable concentration collected post dose. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
h*ng/mL | 6504.88 (2542.12) [lower limit 2542.12] | 8869.21 (2642.17) [lower limit 2642.17]

8. Primary Outcome: Part D: Area Under the Plasma Concentration Time Curve From Time Zero to 24 Hours (AUC[0-24]) for Single Dose of Lazertinib
Description: AUC(0-24) was defined as area under the plasma concentration time curve from time zero to 24 hours. AUC(0-24) for single dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10 and 24 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
h*ng/mL | 3253.58 (916.67) [lower limit 916.67] | 4097.34 (1261.96) [lower limit 1261.96]

9. Primary Outcome: Part D: Maximum Observed Plasma Concentration (Cmax) for Single Dose of Lazertinib
Description: Cmax was defined as maximum observed plasma concentration. Cmax for single dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
Nanograms per milliliter (ng/mL) | 441.04 (135.45) [lower limit 135.45] | 524.13 (271.58) [lower limit 271.58]

10. Primary Outcome: Part D: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Single Dose of Lazertinib
Description: Tmax was defined as time to reach the maximum observed plasma concentration. Tmax for single dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
Hours | 2.00 (0.92) [0.92 to 4.15] | 2.50 (1.07) [1.07 to 4.00]

11. Primary Outcome: Part D: Apparent Terminal Half-Life (t1/2) for Single Dose of Lazertinib
Description: T1/2 was defined the time measured for the plasma concentration of a drug to decrease by half of its initial concentration. T1/2 for single dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
Hours | 51.12 (18.75) [18.75 to 70.71] | 63.98 (52.30) [52.30 to 97.74]

12. Primary Outcome: Part D: Apparent Terminal Elimination Rate Constant (Lambda[z]) for Single Dose of Lazertinib
Description: Lambda(z) was defined as terminal elimination rate constant. Lambda(z) for single dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Per hour (1/h)
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
Per hour (1/h) | 0.02 (0.01) [lower limit 0.01] | 0.01 (0.00) [lower limit 0.00]

13. Primary Outcome: Part D: Apparent Plasma Clearance (CL/F) for Single Dose of Lazertinib
Description: CL/F was defined as apparent plasma clearance. CL/F for single dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters per hour (L/h)
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
Liters per hour (L/h) | 41.92 (15.56) [lower limit 15.56] | 39.38 (12.96) [lower limit 12.96]

14. Primary Outcome: Part D: Apparent Volume of Distribution (Vd/F) for Single Dose of Lazertinib
Description: Vd/F was defined as apparent volume of distribution. Vd/F for single dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
Liters | 2990.36 (1188.45) [lower limit 1188.45] | 3822.19 (984.29) [lower limit 984.29]

15. Primary Outcome: Part D: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the End of Dosing Interval at Steady State (AUCss[0-last]) for Multiple Dose of Lazertinib
Description: AUCss(0-last) was defined as area under the plasma concentration time curve from time zero to end of dosing interval at steady state. AUCss(0-last) for multiple dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose up to 1, 2, 4, 10 and 24 hours post dose on Day 1 of Cycle 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 6
h*ng/mL | 7025.10 (4181.22) [lower limit 4181.22] | 9249.58 (4924.51) [lower limit 4924.51]

16. Primary Outcome: Part D: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) for Multiple Dose of Lazertinib
Description: Cmax,ss was defined as maximum observed plasma concentration at steady state. Cmax,ss for multiple dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose up to 1, 2, 4, 10 and 24 hours post dose on Day 1 of Cycle 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 6
ng/mL | 509.92 (236.66) [lower limit 236.66] | 632.00 (279.88) [lower limit 279.88]

17. Primary Outcome: Part D: Time to Reach Maximum Observed Plasma Concentration at Steady State (Tmax,ss) for Multiple Dose of Lazertinib
Description: Tmax,ss was defined as time to reach maximum observed plasma concentration at steady state. Tmax,ss for multiple dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose up to 1, 2, 4, 10 and 24 hours post dose on Day 1 of Cycle 2
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 6
Hours | 3.15 (1.75) [1.75 to 9.00] | 3.97 (2.22) [2.22 to 9.00]

18. Primary Outcome: Part D: Accumulation Ratio (Rac) for Multiple Dose of Lazertinib
Description: Accumulation ratio was calculated as AUCss(0-last) divided by AUC(0-24), where AUCss(0-last) was defined as area under the plasma concentration time curve from time zero to end of dosing interval at steady state and AUC(0-24) was defined area under the plasma concentration time curve from time zero to 24 hours time. Rac for multiple dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose up to 1, 2, 4, 10 and 24 hours post dose on Day 1 of Cycle 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 11 | 4
Ratio | 2.26 (0.61) [lower limit 0.61] | 2.36 (1.08) [lower limit 1.08]

19. Primary Outcome: Part D: Apparent Plasma Clearance at Steady State (CLss/F) for Multiple Dose of Lazertinib
Description: CLss/F was defined as apparent plasma clearance at steady state. CLss/F for multiple dose of lazertinib was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose up to 1, 2, 4, 10 and 24 hours post dose on Day 1 of Cycle 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters per hour (L/h)
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 6
Liters per hour (L/h) | 44.25 (21.39) [lower limit 21.39] | 50.10 (37.21) [lower limit 37.21]

20. Primary Outcome: Part D: Trough Concentrations (Ctrough) for Multiple Dose of Lazertinib at Cycle 1 Day 1
Description: Ctrough was defined as pre-dose plasma concentration. Ctrough for multiple dose of lazertinib at Cycle 1 Day 1 was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose on Day 1 of Cycle 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
ng/mL | 6.41 (4.55) [lower limit 4.55] | 10.91 (5.99) [lower limit 5.99]

21. Primary Outcome: Part D: Trough Concentrations (Ctrough) for Multiple Dose of Lazertinib at Cycle 1 Day 8
Description: Ctrough was defined as pre-dose plasma concentration. Ctrough for multiple dose of lazertinib at Cycle 1 Day 8 was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose on Day 8 of Cycle 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 14 | 10
ng/mL | 154.62 (87.60) [lower limit 87.60] | 225.47 (168.22) [lower limit 168.22]

22. Primary Outcome: Part D: Trough Concentrations (Ctrough) for Multiple Dose of Lazertinib at Cycle 1 Day 15
Description: Ctrough was defined as pre-dose plasma concentration. Ctrough for multiple dose of lazertinib at Cycle 1 Day 15 was reported in this outcome measure. The concentrations of lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose on Day 15 of Cycle 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
ng/mL | 177.40 (99.23) [lower limit 99.23] | 263.74 (145.61) [lower limit 145.61]

23. Secondary Outcome: Part D: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-last]) of Metabolite M7 After Single Dose of Lazertinib
Description: AUC(0-last) was defined as area under the plasma concentration-time curve from time zero to time of last quantifiable concentration. AUC(0-last) of metabolite M7 after single dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
h*ng/mL | 216.350 (126.357) [lower limit 126.357] | 208.908 (128.968) [lower limit 128.968]

24. Secondary Outcome: Part D: Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC[0-Infinity]) of Metabolite M7 After Single Dose of Lazertinib
Description: AUC(0-infinity) was defined as area under the plasma concentration time curve from time zero to infinite time. AUC(0-infinity) of metabolite M7 after single dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 12 | 7
h*ng/mL | 281.172 (144.163) [lower limit 144.163] | 263.373 (166.254) [lower limit 166.254]

25. Secondary Outcome: Part D: Area Under the Plasma Concentration Time Curve From Time Zero to 24 Hours (AUC[0-24]) of Metabolite M7 After Single Dose of Lazertinib
Description: AUC(0-24) was defined as area under the plasma concentration time curve from time zero to 24 hours. AUC(0-24) of metabolite M7 after single dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10 and 24 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
h*ng/mL | 86.692 (52.492) [lower limit 52.492] | 74.523 (33.137) [lower limit 33.137]

26. Secondary Outcome: Part D: Maximum Observed Plasma Concentration (Cmax) of Metabolite M7 After Single Dose of Lazertinib
Description: Cmax was defined as maximum observed plasma concentration. Cmax of metabolite M7 after single dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
ng/mL | 5.838 (3.946) [lower limit 3.946] | 4.774 (2.257) [lower limit 2.257]

27. Secondary Outcome: Part D: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Metabolite M7 After Single Dose of Lazertinib
Description: Tmax was defined as time to reach the maximum observed plasma concentration. Tmax of metabolite M7 after single dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 9
Hours | 4.020 (2.070) [2.070 to 10.080] | 4.150 (3.080) [3.080 to 22.350]

28. Secondary Outcome: Part D: Apparent Terminal Half-Life (t1/2) of Metabolite M7 After Single Dose of Lazertinib
Description: T1/2 was defined the time measured for the plasma concentration of a drug to decrease by half of its initial concentration. T1/2 of metabolite M7 after single dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 12 | 7
Hours | 41.205 (18.042) [18.042 to 86.989] | 50.019 (13.256) [13.256 to 74.867]

29. Secondary Outcome: Part D: Apparent Terminal Elimination Rate Constant (Lambda [z]) of Metabolite M7 After Single Dose of Lazertinib
Description: Lambda(z) was defined as terminal elimination rate constant. Lambda(z) of metabolite M7 after single dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Per hour (1/h)
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 12 | 7
Per hour (1/h) | 0.017 (0.008) [lower limit 0.008] | 0.021 (0.016) [lower limit 0.016]

30. Secondary Outcome: Part D: Metabolic Ratio (MR) of Metabolite M7 and Lazertinib After Single Dose of Lazertinib
Description: MR was defined as ratio of the AUC(0-infinity) of metabolite M7 and AUC(0-infinity) of lazertinib, where AUC(0-infinity) was defined as area under the plasma concentration time curve from time zero to infinite time. The concentrations of metabolite M7 and lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose, 1, 2, 4, 10, 24 and 48 hours post-dose on Day 1 of Cycle 0
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 12 | 7
Ratio | 0.042 (0.022) [lower limit 0.022] | 0.027 (0.015) [lower limit 0.015]

31. Secondary Outcome: Part D: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the End of Dosing Interval at Steady State (AUCss[0-last]) of Metabolite M7 After Multiple Dose of Lazertinib
Description: AUCss(0-last) was defined as area under the plasma concentration-time curve from time zero to time of the end of dosing interval at steady state. AUCss(0-last) of metabolite M7 after multiple dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose up to 1, 2, 4, 10 and 24 hours post dose on Day 1 of Cycle 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 6
h*ng/mL | 148.335 (89.794) [lower limit 89.794] | 168.765 (159.476) [lower limit 159.476]

32. Secondary Outcome: Part D: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of Metabolite M7 After Multiple Dose of Lazertinib
Description: Cmax,ss was defined as maximum observed plasma concentration at steady state. Cmax,ss of metabolite M7 after multiple dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose up to 1, 2, 4, 10 and 24 hours post dose on Day 1 of Cycle 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 6
ng/mL | 7.866 (4.213) [lower limit 4.213] | 8.319 (7.418) [lower limit 7.418]

33. Secondary Outcome: Part D: Time to Reach Maximum Observed Plasma Concentration at Steady State (Tmax,ss) of Metabolite M7 After Multiple Dose of Lazertinib
Description: Tmax,ss was defined as time to reach the maximum observed plasma concentration at steady state. Tmax,ss of metabolite M7 after multiple dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose up to 1, 2, 4, 10 and 24 hours post dose on Day 1 of Cycle 2
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 6
Hours | 6.330 (2.250) [2.250 to 9.000] | 4.350 (3.930) [3.930 to 24.070]

34. Secondary Outcome: Part D: Accumulation Ratio (Rac) of Metabolite M7 After Multiple Dose of Lazertinib
Description: Accumulation ratio was calculated as AUCss(0-last) divided by AUC(0-24), where AUCss(0-last) was defined as area under the plasma concentration time curve from time zero to end of dosing interval at steady state and AUC(0-24) was defined area under the plasma concentration time curve from time zero to 24 hours. Rac of metabolite M7 after multiple dose of lazertinib was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose up to 1, 2, 4, 10 and 24 hours post dose on Day 1 of Cycle 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 11 | 4
Ratio | 1.976 (0.617) [lower limit 0.617] | 2.270 (1.300) [lower limit 1.300]

35. Secondary Outcome: Part D: Trough Concentrations (Ctrough) of Metabolite M7 After Multiple Dose of Lazertinib at Days 1, 8 and 15 of Cycle 1
Description: Ctrough was defined as pre-dose plasma concentration. Ctrough of Metabolite M7 after multiple dose of lazertinib at Days 1, 8 and 15 of Cycle 1 was reported in this outcome measure. The concentrations of metabolite M7 were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose on Days 1, 8 and 15 of Cycle 1
Population: PK analysis population included all participants who had at least 1 measurable concentration collected post dose. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure. Here 'n' (number analyzed) refers to all participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 14 | 10
ng/mL
  Day 1 Cycle 1: number analyzed (Participants) | 13 | 9
  Day 1 Cycle 1 | 0.257 (0.237) | 0.358 (0.321)
  Day 8 Cycle 1 | 4.928 (3.005) | 5.791 (4.650)
  Day 15 Cycle 1: number analyzed (Participants) | 13 | 9
  Day 15 Cycle 1 | 5.356 (3.604) | 6.340 (4.741)

36. Secondary Outcome: Part D: Metabolic Ratio at Steady State (MRss) of Metabolite M7 and Lazertinib After Multiple Dose of Lazertinib
Description: MRss was defined as ratio of the AUCss(0-last) of metabolite M7 and AUCss(0-last) of lazertinib, where AUCss(0-last) was defined as area under the plasma concentration time curve from time zero to time of end of dosing interval at steady state. The concentrations of metabolite M7 and lazertinib were measured using a validated, specific, and sensitive LC-MS/MS method.
Time Frame: Pre-dose up to 1, 2, 4, 10 and 24 hours post dose on Day 1 of Cycle 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 13 | 6
Ratio | 0.021 (0.006) [lower limit 0.006] | 0.016 (0.009) [lower limit 0.009]

37. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as percentage of participants who had at least 1 confirmed partial or complete response (PR or CR) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 prior to disease progression or recurrence. CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures less than (<) 10 millimeter (mm). PR was defined as greater than or equal to (>=) 30 percent (%) decrease in sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-progressive disease (PD). PD was defined as >=20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative 20% increase, sum must also demonstrate an absolute increase of >=5 mm. Appearance of one or more new lesions was considered progression.
Time Frame: Up to 33.7 months
Population: Evaluable for response population included all participants in safety analysis population who had a baseline RECIST version 1.1 assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 15 | 13
Percentage of participants | 26.7 (4.3) [4.3 to 49.0] | 7.7 (0.0) [0.0 to 22.2]

38. Secondary Outcome: Duration of Response (DoR)
Description: DOR was defined as time between date of first documented confirmed response (PR/CR) and date of first documented progression or death, whichever occurred first. CR was defined as disappearance of target and non-target lesions and normalization of tumour markers. Pathological lymph nodes short axis measures <10 mm. PR was defined as >=30% decrease in sum of measures (tumour lesions-longest diameter and nodes-short axis)of target lesions, taking as reference baseline sum of diameters. PD was defined as >=20% increase in sum of diameters of measured lesions taking as references smallest sum of diameters recorded on study(including baseline), absolute increase of >=5 mm/appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions.
Time Frame: Up to 33.7 months
Population: Evaluable for response population included all participants in safety analysis population who had a baseline RECIST version 1.1 assessment. Here 'N' (number of participants analyzed) refers to number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 4 | 1
Months | NA [5.6 to NA] — Due to low sample size, median was not reached and upper limit of 95% confidence interval (CI) could not be calculated. | 2.8 [NA to NA] — Due to low sample size, lower and upper limit of 95% CI could not be calculated.

39. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as percentage of participants with a best overall response (BOR), extracranial and intracranial response of CR, PR or stable disease (SD). As per RECIST version 1.1 CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. PR was defined as >=30% decrease in sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference baseline sum of diameters. Non-target lesions must be non-PD. PD was defined as >=20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to relative 20% increase, sum must also demonstrate >=5 mm absolute increase. Appearance of one or more new lesions was considered progression. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to 33.7 months
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 15 | 13
Percentage of participants | 60.0 (35.2) [35.2 to 84.8] | 53.8 (26.7) [26.7 to 80.9]

40. Secondary Outcome: Percentage Change From Baseline in Tumor Size
Description: Tumor size was defined as the sum lengths of the longest diameters of the target lesion. Percentage change in tumor size was determined for participants with measurable disease at baseline. Baseline for RECIST version 1.1 was defined as the last evaluable assessment prior to starting treatment.
Time Frame: Baseline up to 33.7 months
Population: Evaluable for response population included all participants in safety analysis population who had a baseline RECIST version 1.1 assessment. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change in tumor size
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 14 | 12
Percentage change in tumor size | -5.37 (37.68) [lower limit 37.68] | 9.56 (42.89) [lower limit 42.89]

41. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of first dose of study drug to the earliest date of disease progression per RECIST version 1.1, or death due to any cause, whichever occurs first. PD was defined as at least 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) and an absolute increase of >=5 mm or appearance of at least 1 new lesion.
Time Frame: Up to 33.7 months
Population: The safety analysis population included all participants who received at least 1 dose of IP. Here 'N' (number of participants analyzed) refers to the number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 11 | 11
Months | 3.1 (1.3) [1.3 to 11.2] | 4.2 (0.0) [0.0 to 7.7]

42. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose to date of death due to any cause.
Time Frame: Up to 33.7 months
Population: as for outcome 41
Measure: Median (Full Range); unit: Months
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
Number analyzed (Participants) | 11 | 9
Months | 9.1 (2.6) [2.6 to 24.3] | 7.7 (3.4) [3.4 to 12.3]

ADVERSE EVENTS:
Time Frame: All cause mortality: Day 1 up to 33.7 months; Serious and other adverse events: Day 1 up to 32.7 months
Description: The safety analysis population included all participants who received at least 1 dose of investigational product (IP).
Arm/Group | Lazertinib 240 mg | Lazertinib 320 mg
All-Cause Mortality (participants affected / at risk) | 11/15 | 9/13
Serious Adverse Events (participants affected / at risk) | 10/15 | 6/13
Other Adverse Events (participants affected / at risk) | 15/15 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lazertinib 240 mg (N=15) | Lazertinib 320 mg (N=13)
Palpitations (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Pain (General disorders) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Adrenalectomy (Surgical and medical procedures) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lazertinib 240 mg (N=15) | Lazertinib 320 mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 7 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0
Dry Eye (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 7
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gingival Pain (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 8
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 3 | 2
Chest Pain (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 3
Gait Disturbance (General disorders) | 1 | 1
Induration (General disorders) | 1 | 0
Medical Device Pain (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 3 | 2
Pain (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Covid-19 (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 3 | 2
Amylase Increased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 4 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 2 | 3
Blood Magnesium Decreased (Investigations) | 1 | 0
Blood Sodium Decreased (Investigations) | 1 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 3 | 0
Platelet Count Decreased (Investigations) | 0 | 1
Troponin I Increased (Investigations) | 1 | 1
Troponin Increased (Investigations) | 1 | 1
Weight Decreased (Investigations) | 1 | 1
White Blood Cell Count Decreased (Investigations) | 1 | 1
Appetite Disorder (Metabolism and nutrition disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 1
Memory Impairment (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Taste Disorder (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Affect Lability (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Depressed Mood (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Sleep Disorder (Psychiatric disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Paronychia (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 3
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Solar Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hot Flush (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study Parts A, B, and C were sponsored by Yuhan Corporation under protocol identifier (ID) YH25448-201 and Part D was sponsored by Janssen Research and Development, LLC under protocol ID 73841937NSC2001. Therefore, only Part D results are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All draft publications, including abstracts or detailed summaries of any proposed presentations, must be submitted to the Sponsor at the earliest practicable time for review, but in any event not less than 30 days before submission or presentation unless otherwise set forth in the clinical trial agreement (CTA).

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT04075396/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT04075396/SAP_001.pdf